CLINICAL TRIAL: NCT00319319
Title: A Double-Blind,Randomized,Placebo-Controlled Trial of Mecamylamine Hydrochloride for the Treatment of SSRI-Refractory Major Depressive Disorder.
Brief Title: Nicotinic Receptor Augmentation of SSRI Antidepressants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF-02-006
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Depressive Disorder
Keywords: major depressive disorder,; serotonin selective reuptake inhibitor,; mecamylamine,; controlled trial,; cigarette smoking
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Cigarette Smoking | interventions — Mecamylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mecamylamine hydrochloride (Inversine)

SUMMARY:
The purpose of this study is to determine whether the nicotinic receptor antagonist mecamylamine hydrochloride (Inversine) can augment SSRI-refractory major depression symptoms, quality of life and cigarette smoking outcomes. A total of n=60 SSRI-refractory patients who are on stable doses of an SSRI are being recruited into this 8-week double-blind, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
Mecamylamine for the Treatment of Depression in SSRI-Treated Partial Responders

A. Purpose

1. To compare the nicotinic receptor antagonist mecamylamine (MEC) to placebo for the treatment of depressive symptoms in nicotine-dependent, cigarette smokers and in non-smokers who are maintained on, and are partial responders to serotonin-selective reuptake inhibitors (SSRIs).
2. To determine the effects of MEC versus placebo on cigarette smoking behavior in SSRI-maintained depressed smokers and non-smokers.

B. Background The co-morbid rates of nicotine dependence in patients with major depression are estimated to be 50-60% [1-3]. Smokers with a history of major depression disorders have great difficulty quitting smoking compared to smokers without a history of major depression [2, 4]. Furthermore, smokers with a history of depression appear to be at substantial risk for the emergence of depressive symptom exacerbation, typically within one month after smoking cessation [2, 5-7], though this phenomenon has been recently questioned [8]. Recent estimates are that nearly 45% of all cigarettes consumed in the USA are by individuals with mental illness [10].

These clinical relationships between tobacco use and depression do suggest some important effects of nicotine and nicotinic receptor mechanisms in major depressive disorder. Thus, it has been postulated that nicotine and cigarette smoking may exert antidepressant effects [4, 5, 11, 12], presumably mediated through stimulation of nicotinic acetylcholine receptor (nAChR) systems. In fact, it has been shown in an open-label trial that nicotine patch could produce substantial antidepressant effects with 3 days of transdermal nicotine administration in non-smoking subjects with major depression [12].

Based on the results of several studies, serotonin-selective reuptake inhibitors (SSRIs) have not shown promise as anti-smoking pharmacotherapies [5, 9]. However, bupropion and several SSRIs (including fluoxetine, sertraline, fluvoxamine and paroxetine) have been shown using in vitro studies to bind, at clinically relevant concentrations, to the non-competitive ion channel site of the high-affinity nAChR [11], the same site to which mecamylamine (MEC) binds. Since MEC has been shown to have mood-enhancing effects in a controlled smoking cessation study examining the combination of MEC and NTP [13], and recently to have mood-stabilizing properties in patients with bipolar symptoms [14], we speculate that the combination of MEC with an SSRI may have significant positive effects on both depressive symptoms and smoking. In on-going work at Yale using transgenic mice with deletion of the alpha 2-subunit of the nAChR, Picciotto and colleagues have demonstrated that the antidepressant effects of the tricyclic antidepressant amitriptyline in a learned helplessness model of depression are abolished in alpha 2-subunit knock-out mice (which lack functional high-affinity nAChRs containing the alpha 2-subunit) compared to the control background (C57B/L) mouse strain (M.R. Picciotto, Ph.D., personal communication). This finding suggests that the presence of functional nAChRs is necessary, but not sufficient, for generation of antidepressant responses to amitriptyline, an antidepressant that has also been shown to non-competitively inhibit high-affinity nAChRs [11]. Thus, since both SSRIs and MEC bind to nAChRs and since nAChRs may mediate the effects of most clinically effective of antidepressants, it is possible that the combination of MEC with an SSRI may serve to augment partial antidepressant responses to SSRIs, and reduce the drive to smoke in these patients, either primarily or secondarily.

The current study proposes to evaluate the nicotinic receptor antagonist mecamylamine (Inversine®) in comparison to matching placebo, in the treatment of depressive symptoms in smokers and non-smokers with major depressive disorder. These subjects would be maintained on antidepressant treatment with serotonin-selective reuptake inhibitors, and continue to exhibit at least mild depressive symptoms (e.g. partial antidepressant responders). The primary outcome measure will be depressive symptoms at the end of the 12-week trial (e.g. a 50% decrease in depressive symptoms) compared to baseline. Furthermore, we will compare the effects of mecamylamine versus placebo on smoking behavior in these SSRI-maintained partial responders.

C. Specific Location of Study: The study will be conducted at the Program for Research in Smokers with Mental Illness (PRISM), Substance Abuse Center, Connecticut Mental Health Center (CMHC), New Haven, CT.

D. Probable Duration of Project - (3/1/02-12/31/06)

E. Research Plan and Data and Safety Monitoring Plan Study Medication: Mecamylamine hydrochloride has been on the market since 2000 and is FDA approved for the treatment of hypertension. Mecamylamine HCI is currently made by Targacept, Inc. We will purchase Mecamylamine study medication through local pharmacies and the CMHC pharmacist will make placebo capsules.

Inclusion Criteria:

1. Have a history of major depression based on SCID, and currently maintained on an SSRI antidepressant with no dose changes in the past three months.
2. May have a history of bipolar disorder, with no evidence of manic or hypomanic episode in the past year and currently in depressive phase of Bipolar I or II disorder.
3. May have a history of depression with psychotic features with no current evidence of psychotic features in the past year and not currently treated with an antipsychotic medication.
4. Current depressive symptoms will be assessed to be mild to moderate, and Beck Depression Inventory scores of 10-30.
5. Capable of giving informed consent.
6. For smoking subjects, meet DSM-IV criteria for nicotine dependence, smoking at least 15 cigarettes/day, biochemically verified.
7. For smoking subjects, no intention to quit smoking.
8. Adults age 18-65.

Exclusion Criteria:

1. A history of alcohol or drug dependence or abuse in the six months prior to study entry.
2. A history of schizophrenia or schizoaffective disorder, or currently treated with antipsychotic medications.
3. A history of a manic or psychotic episode within the past year.
4. Currently treated with antidepressants other than SSRIs.
5. Presence of suicidal or homicidal ideation at the time of study entry, and/or evidence of significant impairment in functioning that would necessitate treatment of the subject in a non-outpatient setting.
6. If female, currently pregnant (as assessed by urine pregnancy test at baseline and as appropriate thereafter), or planning to become pregnant during the course of the trial. 7) Current history of glaucoma (open- and closed angle), prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis and pyloric stenosis..

8) A history of hypotension (e.g. systolic blood pressure less than 90mm Hg). 9) A history of known contraindications to Mecamylamine (Inversine) 10) For smokers, currently taking bupropion (either Wellbutrin or Zyban preparations) or nicotine replacement therapies, or currently involved in smoking cessation behavioral therapies.

Study Design:

Subjects who have a history of major depression partially responsive to an SSRI and either dependent cigarette smokers (N=30) or non-smokers (N=30) will be recruited into this study. The study design is a 2 (smoking status) x 2 (study medication) configuration for 8 weeks.

Treatments Groups:

Smoker Subjects:

1. Placebo (Placebo tablets, one po bid, N=15)
2. Mecamylamine (10.0 mg/day as 5 mg po bid; N=15)

   Non-Smoker Subjects:
3. Placebo (Placebo tablets, one po bid, N=15)
4. Mecamylamine (10.0 mg/day; as 5.0 mg po bid, N=15)

Subjects will begin MEC in Week 2 at 0.0/5.0 mg qd (2 tablets po qd), which will be increased to 0.0/5.0 mg po bid (2 tablets po bid) during Day 8 of the trial (Week 2). Study medications will be continued until the end of Week 8. If the subject finds the study medication, mecamylamine, to be helpful, this information can be shared with the subject's physician to enable a decision about whether mecamylamine should be continued after the study, since it is available by prescription from the subject's physician. Both smoker and non-smoker participants would receive supportive therapy intervention for the treatment.

G. Economic Considerations:

Subjects would be paid $25.00 for completion of baseline assessments and $25.00 for successful completion of the 8-week trial. Thus, subjects could earn up to $50.00 for their study participation.

III. HUMAN SUBJECTS A. Subject Population, Recruitment: A total of 60 smoking (n=30) and non-smoking (n=30) subjects with current depressed and treated with a serotonin-selective reuptake inhibitor (SSRI) will be recruited.

B. Source of Research Material: Study medication (Mecamylamine 2.5 mg) will be purchased from local pharmacies. Placebo medication will be prepared by CMHC pharmacist using encapsulation.

C. Consent Procedures: Subjects will be recruited for participation and provided with a written consent form requiring their signature. Only subjects capable of giving informed consent and scoring 80% on post-consent test will be admitted into the study.

D. Risks: The primary risks in this study are those associated with the study medication, mecamylamine. Side effects associated with mecamylamine include constipation, dry mouth, nausea and vomiting, orthostatic hypotension (dizziness when standing) and, very rarely, unusual muscle movements and seizures. In our experience, constipation appears to be the most common side effect.

Because the study medication, mecamylamine, may cause a drop in blood pressure, we plan to monitor each subject's blood pressure (sitting and standing) on a weekly basis. If a subject develops a systolic blood pressure < 100mm Hg, we will plan to monitor blood pressure twice weekly. If a subject develops a systolic blood <90mm Hg, we will plan to discontinue study medication. Lastly, if a subject experiences a systolic blood pressure drop >10mm Hg, we will plan to monitor twice weekly or until the problems resolves.

In addition, we will exclude potential subjects with a history of glaucoma, prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis, pyloric stenosis, and a history of hypersensitivity to mecamylamine. There is the rare chance that if a smoking subject quit smoking during this study, the subject could have a worsening of depressive symptoms.

E. Protection of Subjects: All reports generated from the data obtained through this study will protect the confidentiality of the subjects who participate in this study. In case of a medical emergency, the medication group blinding can be broken by the principal investigator. If a depressed subject shows clinical deterioration, Dr. George and Ms. Vessicchio will determine: 1) whether subject can remain in the study, or; 2) whether a higher level of care is needed.

G. Confidentiality: All reports generated from this study will not contain any identifying information about the participants.

ELIGIBILITY:
Inclusion Criteria:

* Major depression, recurrent outpatients, ages 18-65, smoker or non-smoker, on SSRI monotherapy, depression scores on HDRS-17 item scale or = 12.

Exclusion Criteria:

* suicidal or homicidal ideation, need for inpatient or partial hospital care, systolic blood pressure <100 mm Hg, history of hypersensitivity to mecamylamine or its excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale
Beck Depression Inventory

SECONDARY OUTCOMES:
Cigarette Smoking
Quality of Life
Clinical Global Impression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Tony P. George, M.D., Principal Investigator — Yale University School of Medicine, Psychiatry
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] George TP, Sacco KA, Vessicchio JC, Weinberger AH, Shytle RD. Nicotinic antagonist augmentation of selective serotonin reuptake inhibitor-refractory major depressive disorder: a preliminary study. J Clin Psychopharmacol. 2008 Jun;28(3):340-4. doi: 10.1097/JCP.0b013e318172b49e. PMID 18480694